CLINICAL TRIAL: NCT02720614
Title: A Phase II Study of Accelerated Hypofractionated Three-dimensional Conformal Radiation Therapy Concurrent With Chemotherapy in Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: Hypofractionated Radiation Therapy Combined With Concurrent Chemotherapy for Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LIN QIANG (Other)
Responsible Party: Sponsor-Investigator, LIN QIANG, Professor, North China Petroleum Bureau General Hospital
Organization: North China Petroleum Bureau General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NorthChinaPBGH
Record Dates: First submitted 2016-03-23; First posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: accelerated hypofractionated radiotherapy; three-dimensional conformal radiation therapy; concurrent radiochemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypofractionated radiation/chemotherapy (Experimental): Hypofractionated radiation：Patients receive accelerated hypofractionated radiation: three-dimensional conformal radiation therapy (3-DCRT) with a total dose of 69 Gy, delivered at 3 Gy per fraction, once daily, five fractions per week, completed within 4.6 weeks.
  Chemotherapy: Regimen 1 is as follows: vinorelbine (NVB) was administered by intravenous infusion at a dose of 25 mg/m2 on day 1 (d1) and day 8 (d8), and carboplatin (CBP) is administered at a concentration-time curve (AUC) of 5 mg/ml on d8. This treatment was repeated every 28 days. One cycle of chemotherapy is performed concurrently with the radiotherapy.
  Chemotherapy: Regimen 2 is as follows: paclitaxel at 30 mg/m2 and cisplatin at 20 mg/m2 (TP) are administrated every week for 5 weeks continuously.
  Interventions: Radiation: Hypofractionated radiation/chemotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiation/chemotherapy — Procedure: Radiation Therapy Drug: Vinorelbine Drug: Carboplatin Drug: Paclitaxel Drug: Cisplatin

SUMMARY:
The purpose of this study is to evaluate the safety of accelerated hypofractionated three-dimensional conformal radiation therapy (3 Gy/fraction) concurrent with chemotherapy for patients with unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
Increasing the biological effective dose (BED) of radiotherapy for non-small cell lung cancer (NSCLC) can increase local control rates and improve overall survival. Compared with conventional fractionated radiotherapy, accelerated hypofractionated radiotherapy can yield higher BED, shorten the total treatment time, and theoretically obtain better efficacy. However, currently, there is no optimal hypofractionated radiotherapy regimen. Based on phase I trial results, we performed this phase II trial to further evaluate the safety and preliminary efficacy of accelerated hypofractionated three-dimensional conformal radiation therapy(3-DCRT) combined with concurrent chemotherapy for patients with unresectable stage III NSCLC.

Patients with previously untreated unresectable stage III NSCLC received 3-DCRT with a total dose of 69 Gy, delivered at 3 Gy per fraction, once daily, five fractions per week, completed within 4.6 weeks. At the same time, platinum doublet chemotherapy was applied.

ELIGIBILITY:
Inclusion Criteria:

* Pathological or cytological diagnose of unresectable stage III non-small cell lung cancer
* The Karnofsky performance status (KPS) score ≥70.
* The expected survival time ≥3 months.
* Adequate blood, liver, lungs and kidney function
* Accessible contact information
* Informed consent required before enrollment.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Another malignant tumor history (with the exception of patients with cervical carcinoma in situ and non-malignant melanoma skin cancer that had been clinically cured for at least 5 years)
* Cannot receive concurrent chemotherapy due to medical reasons.
* Superior vena cava syndrome.
* Severe lung diseases that affected lung function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Severe and Life-threatening Adverse Events (AE) | Baseline to the time of intolerable toxicity(up to 1 year) or measured Progressive Disease (PD)
  intolerable toxicities: severe and life-threatening adverse events (Grade III/IV in Common Terminology Criteria for Adverse Events v3.0 (CTCAE 3.0))

SECONDARY OUTCOMES:
Percentage of Participants with Progression Free Survival (PFS) at 1 Year | Baseline and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lin, Dr, Study Chair — North China Petroleum Bureau General Hospital of Hebei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Chen W, Zheng R, Zhang S, Zhao P, Zeng H, Zou X. Report of cancer incidence and mortality in China, 2010. Ann Transl Med. 2014 Jul;2(7):61. doi: 10.3978/j.issn.2305-5839.2014.04.05. PMID 25333036
- [Background] Bayman N, Blackhall F, McCloskey P, Taylor P, Faivre-Finn C. How can we optimise concurrent chemoradiotherapy for inoperable stage III non-small cell lung cancer? Lung Cancer. 2014 Feb;83(2):117-25. doi: 10.1016/j.lungcan.2013.11.017. Epub 2013 Dec 1. PMID 24373738
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Lin Q, Liu YE, Ren XC, Wang N, Chen XJ, Wang DY, Zong J, Peng Y, Guo ZJ, Hu J. Dose escalation of accelerated hypofractionated three-dimensional conformal radiotherapy (at 3 Gy/fraction) with concurrent vinorelbine and carboplatin chemotherapy in unresectable stage III non-small-cell lung cancer: a phase I trial. Radiat Oncol. 2013 Aug 17;8(1):201. doi: 10.1186/1748-717X-8-201. PMID 23957889
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Koukourakis M, Hlouverakis G, Kosma L, Skarlatos J, Damilakis J, Giatromanolaki A, Yannakakis D. The impact of overall treatment time on the results of radiotherapy for nonsmall cell lung carcinoma. Int J Radiat Oncol Biol Phys. 1996 Jan 15;34(2):315-22. doi: 10.1016/0360-3016(95)02102-7. PMID 8567332
- [Background] Beli I, Koukourakis G, Platoni K, Tolia M, Kelekis N, Kouvaris J, Syrigos C, Mystakidou K, Varveris C, Kouloulias V. Hypofractionated radiotherapy in non small cell lung cancer: a review of the current literature. Rev Recent Clin Trials. 2010 May;5(2):103-11. doi: 10.2174/157488710791233608. PMID 20423316
- [Background] Oh D, Ahn YC, Kim B, Pyo H. Hypofractionated three-dimensional conformal radiation therapy alone for centrally located cT1-3N0 non-small-cell lung cancer. J Thorac Oncol. 2013 May;8(5):624-9. doi: 10.1097/JTO.0b013e31828cb6db. PMID 23584294
- [Background] Faria SL, Souhami L, Portelance L, Duclos M, Vuong T, Small D, Freeman CR. Absence of toxicity with hypofractionated 3-dimensional radiation therapy for inoperable, early stage non-small cell lung cancer. Radiat Oncol. 2006 Nov 1;1:42. doi: 10.1186/1748-717X-1-42. PMID 17078878
- [Background] Amini A, Lin SH, Wei C, Allen P, Cox JD, Komaki R. Accelerated hypofractionated radiation therapy compared to conventionally fractionated radiation therapy for the treatment of inoperable non-small cell lung cancer. Radiat Oncol. 2012 Mar 15;7:33. doi: 10.1186/1748-717X-7-33. PMID 22420631
- [Background] McPartlin AJ, Chaudhry S, Swindell R, Bayman N, Burt P, Chittalia A, Cootes J, Faivre Finn C, Harris M, Lander H, Lee L, Sheikh H, Pemberton L. The largest UK single centre series using hypofractionated radical radiotherapy for NSCLC in the very elderly. Lung Cancer. 2013 Jul;81(1):144. doi: 10.1016/j.lungcan.2013.03.010. Epub 2013 May 2. No abstract available. PMID 23643277
- [Background] Bral S, Duchateau M, Versmessen H, Engels B, Tournel K, Vinh-Hung V, De Ridder M, Schallier D, Storme G. Toxicity and outcome results of a class solution with moderately hypofractionated radiotherapy in inoperable Stage III non-small cell lung cancer using helical tomotherapy. Int J Radiat Oncol Biol Phys. 2010 Aug 1;77(5):1352-9. doi: 10.1016/j.ijrobp.2009.06.075. Epub 2010 Jan 7. PMID 20056350
- [Background] Tho LM, Mahmood R, Leitch M, Brisbane I, Kakumanu S, Mohammed N. Oesophageal toxicity and hypofractionated concurrent chemoradiotherapy for non-small cell lung cancer. Clin Oncol (R Coll Radiol). 2009 Feb;21(1):74. doi: 10.1016/j.clon.2008.10.003. Epub 2008 Nov 5. No abstract available. PMID 18986800
- [Background] Maguire J, Khan I, McMenemin R, O'Rourke N, McNee S, Kelly V, Peedell C, Snee M. SOCCAR: A randomised phase II trial comparing sequential versus concurrent chemotherapy and radical hypofractionated radiotherapy in patients with inoperable stage III Non-Small Cell Lung Cancer and good performance status. Eur J Cancer. 2014 Nov;50(17):2939-49. doi: 10.1016/j.ejca.2014.07.009. Epub 2014 Oct 7. PMID 25304298
- [Background] Kim JO, Chu KP, Fairchild A, Ghosh S, Butts C, Chu Q, Gabos Z, Joy AA, Nijjar T, Robinson DM, Sangha R, Scrimger R, Smylie M, Yee D, Roa WH. Dose-escalated Hypofractionated Intensity-modulated Radiation Therapy With Concurrent Chemotherapy for Inoperable or Unresectable Non-Small Cell Lung Cancer. Am J Clin Oncol. 2017 Jun;40(3):294-299. doi: 10.1097/COC.0000000000000140. PMID 25333733
- [Background] Koukourakis MI, Patlakas G, Froudarakis ME, Kyrgias G, Skarlatos J, Abatzoglou I, Bougioukas G, Bouros D. Hypofractionated accelerated radiochemotherapy with cytoprotection (Chemo-HypoARC) for inoperable non-small cell lung carcinoma. Anticancer Res. 2007 Sep-Oct;27(5B):3625-31. PMID 17972527
- [Background] Belderbos J, Uitterhoeve L, van Zandwijk N, Belderbos H, Rodrigus P, van de Vaart P, Price A, van Walree N, Legrand C, Dussenne S, Bartelink H, Giaccone G, Koning C; EORTC LCG and RT Group. Randomised trial of sequential versus concurrent chemo-radiotherapy in patients with inoperable non-small cell lung cancer (EORTC 08972-22973). Eur J Cancer. 2007 Jan;43(1):114-21. doi: 10.1016/j.ejca.2006.09.005. Epub 2006 Nov 3. PMID 17084621
- [Background] Bearz A, Minatel E, Rumeileh IA, Borsatti E, Talamini R, Franchin G, Gobitti C, Del Conte A, Trovo M, Baresic T. Concurrent chemoradiotherapy with tomotherapy in locally advanced Non-Small Cell Lung Cancer: a phase I, docetaxel dose-escalation study, with hypofractionated radiation regimen. BMC Cancer. 2013 Oct 31;13:513. doi: 10.1186/1471-2407-13-513. PMID 24176164
- [Background] Matsuura K, Kimura T, Kashiwado K, Fujita K, Akagi Y, Yuki S, Murakami Y, Wadasaki K, Monzen Y, Ito A, Kagemoto M, Mori M, Ito K, Nagata Y. Results of a preliminary study using hypofractionated involved-field radiation therapy and concurrent carboplatin/paclitaxel in the treatment of locally advanced non-small-cell lung cancer. Int J Clin Oncol. 2009 Oct;14(5):408-15. doi: 10.1007/s10147-009-0889-0. Epub 2009 Oct 25. PMID 19856048
- [Background] Ohri N, Dicker AP, Lawrence YR. Can drugs enhance hypofractionated radiotherapy? A novel method of modeling radiosensitization using in vitro data. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):385-93. doi: 10.1016/j.ijrobp.2011.06.1990. Epub 2012 Jan 19. PMID 22265460
- [Background] Zhu ZF, Fan M, Wu KL, Zhao KL, Yang HJ, Chen GY, Jiang GL, Wang LJ, Zhao S, Fu XL. A phase II trial of accelerated hypofractionated three-dimensional conformal radiation therapy in locally advanced non-small cell lung cancer. Radiother Oncol. 2011 Mar;98(3):304-8. doi: 10.1016/j.radonc.2011.01.022. Epub 2011 Feb 21. PMID 21345508
- [Derived] Ren XC, Wang QY, Zhang R, Chen XJ, Wang N, Liu YE, Zong J, Guo ZJ, Wang DY, Lin Q. Accelerated hypofractionated three-dimensional conformal radiation therapy (3 Gy/fraction) combined with concurrent chemotherapy for patients with unresectable stage III non-small cell lung cancer: preliminary results of an early terminated phase II trial. BMC Cancer. 2016 Apr 23;16:288. doi: 10.1186/s12885-016-2314-1. PMID 27108080